CLINICAL TRIAL: NCT06684431
Title: A Phase I Study to Evaluate Safety and Immunogenicity of DNA Vaccine N-pVAX1 Against Crimean Congo Hemorrhagic Fever
Brief Title: Study to Evaluate Safety and Immunogenicity of DNA Vaccine N-pVAX1 Against Crimean Congo Hemorrhagic Fever
Acronym: CCHF-NP-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Matti Sällberg, Director of Department of Laboratory Medicine, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCHF-NP-1
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Crimean Congo Hemorrhagic Fever
Keywords: N-pVAX1; Phase I; Dose-escalation
MeSH Terms: conditions — Hemorrhagic Fever, Crimean

STUDY DESIGN:
Intervention Model Description: Dose-escalation: first low-dose group (n=5), then mid-dose group (n=5), last high-dose group (n=5)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine (Experimental): N-pVAX1 vaccine
  Interventions: Biological: N-pVAX1

INTERVENTIONS:
Biological: N-pVAX1 — Crimean Congo Hemorrhagic Fever Vaccine

SUMMARY:
This First-in-human dose-escalation vaccine phase I study aims to evaluate safety and reactogenicity of the investigational vaccine N-pVAX1, against Crimean Congo Hemorrhagic Fever, delivered by in vivo EP given as three im doses at weeks 0, 4 and 12.

DETAILED DESCRIPTION:
This First-in-human dose-escalation vaccine phase I study aims to evaluate safety and reactogenicity of the investigational vaccine N-pVAX1, against Crimean Congo Hemorrhagic Fever, delivered by in vivo EP given as three im doses at weeks 0, 4 and 12.

The study vaccine dose is planned to be staggered, starting with the low-dose group (0.45 mg), followed by the mid-dose group (0.9 mg), and finally the high-dose group (1.8 mg). In total 15 healthy volunteers at the ages of 18-60 will be enrolled.

Primary objective:

• The primary objective of this study is to assess the safety and reactogenicity of the investigational vaccine N-pVAX1 delivered by in vivo EP given as three im doses at weeks 0, 4 and 12.

The secondary objectives:

• To investigate the humoral immune response to the investigational vaccine administered as three doses, by measuring CCHF nucleocapsid antibody levels.

Exploratory objective:

• To investigate in more detail the humoral response and to analyze the cellular immune response to the investigational vaccine.

Trial participants will be followed-up for local and systemic adverse reactions throughout the study period. Blood samples to measure presence of antibody levels to the vaccine components and cellular immunity will be taken at Day 14 and 28 post first and second vaccine dose and at Day 14 and 3 months post last vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 60 years (at the time of consent).
2. Healthy participant, according to the investigator's clinical judgment, as established by medical history, vital signs, physical examination, and laboratory assessments.
3. No clinically significant laboratory abnormalities as determined by the investigator at screening.

   Note: one retest of lab tests is allowed within the screening window.
4. Negative HIV 1/2 antibody/antigen test, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody at screening.
5. Participant with a body mass index (BMI) 20-30.0 kg/m2.
6. Provide written informed consent before initiation of any study procedures.
7. A female participant is eligible for this study if she is one of the following:

   * of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year)
   * of childbearing potential but agrees to practice highly effective contraception or abstinence (if this is the preferred and usual lifestyle of the participant) from 30 days prior to vaccination up to 3 months after last vaccination.

   Highly effective methods of contraception include one or more of the following:
   1. male partner who is sterile (vasectomised) prior to the female study subject's entry into the study and is the sole sexual partner for the female subject;
   2. hormonal (oral, intravaginal, transdermal, implantable or injectable)
   3. an intrauterine hormone-releasing system (IUS)
   4. an intrauterine device (IUD) with a documented failure rate of < 1%.
8. A female participant is eligible if she is willing to abstain from donating oocyte and a male participant if he is willing to abstain from donating sperm from the screening visit up to 3 months after last vaccination.
9. A male participant who is sexually active is eligible if he is willing to use a condom from the screening visit up to 3 months after last vaccination except if the male participant is sterile (e.g. vasectomised); the unique female sexual partner is postmenopausal, is permanently sterilized (e.g. hysterectomy or tubal ligation), or use a highly effective method of contraception.
10. Able to understand and comply with planned study procedures and willing to be available for all study-required procedures, visits and calls for the duration of the study.

Exclusion Criteria:

1. History of presence of pulmonary disorders (chronic obstructive pulmonary lung disease etc) or asthma (exception of allergic asthma, which is allowed).
2. History or presence of thrombocytopenia and/or bleeding disorders.
3. A positive serum pregnancy test at screening or urine pregnancy test prior to study injection, women who are planning to become pregnant during the study, or women who are breastfeeding.
4. Clinically relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, inflammatory, autoimmune, central nervous system or neurological diseases.
5. Use of immunosuppressive drugs as e.g. corticosteroids (excluding topical preparations and inhalers) within 3 months prior to vaccination or 6 months for chemotherapies and all along the study.
6. Vaccination within 2 weeks prior to vaccination or planning to receive a licensed vaccine before month 3 (e.g. inactivated influenza vaccine).
7. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of known or suspected allergic reaction likely to be exacerbated by any component of the Investigational vaccine.
8. Participation in another investigational clinical study within four weeks before the screening visit or planned before the study completion.
9. Subjects with confirmed or suspected immunodeficiency.
10. Any condition that in the opinion of the principal investigator (PI) would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Local reactions | For up to 7 days after each vaccine dose
  Local reactions (pain at the injection site, redness, and swelling) for up to 7 days after each vaccine dose.
Visual analogue scale (VAS) score | At vaccination (0 minutes), and after 5, 15, 30 and 60 minutes post-EP
  Visual analogue scale (VAS) score to rate the level of pain experienced immediately (0 minutes), and after 5, 15, 30 and 60 minutes post-EP.
Systemic events | For 7 days after each vaccine dose
  Systemic events (fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain) for 7 days after each vaccine dose.
Unsolicited AEs | From the first study dose to 28 days after the last vaccination
  Unsolicited AEs from the first study dose to 28 days after the last vaccination.
Serious Adverse Events (SAEs)/suspected unexpected serious adverse reactions (SUSARs) | From the first study dose until the study end at 3 months after last vaccination
  Serious Adverse Events (SAEs)/suspected unexpected serious adverse reactions (SUSARs) from the first study dose until the study end at 3 months after last vaccination.

SECONDARY OUTCOMES:
Change in antibody levels to the CCHF nucleocapsid protein | At Baseline, day 14 and 28 post vaccine dose and at 3 months post last vaccine dose
  Change from baseline sample (a two-fold increase in endpoint titer or a 50% increase in optical density at a 1:62, 1:125, 1:250, 1:500, or 1:1000 serum dilution) in antibody levels to the CCHF nucleocapsid protein by inhouse and/or commercial assays during the study period.

OTHER OUTCOMES:
Exploratory: Description of in depth humoral and cellular immunological responses | At Baseline, day 14 and 28 post vaccine dose and at 3 months post last vaccine dose
  Description of in depth humoral and cellular immunological responses after receiving investigational vaccine at each sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Aleman, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Phase I Unit, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No